CLINICAL TRIAL: NCT05069220
Title: A Study of 18F-MFBG Imaging for the Tumor Burden Evaluation or Diagnostic Performance in Pheochromocytoma, Paraganglioma and Neuroblastoma.
Brief Title: 18F-MFBG PET/CT in the Evaluation of Neural Crest Tumor
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZS-3060MFBG
Record Dates: First submitted 2021-09-20; First posted 2021-10-06 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Neuroendocrine Tumor; Neuroblastoma; Pheochromocytoma; Paraganglioma
MeSH Terms: conditions — Neuroendocrine Tumors; Neuroblastoma; Pheochromocytoma; Paraganglioma | interventions — 3-fluorobenzylguanidine; gallium Ga 68 dotatate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-MFBG PET/CT in neuroendocrine malignancies (Experimental): Each patient receive a single intravenous injection of 18F-MFBG 2-4 MBq/kg and undergo PET/CT scan after 60 min post-injection. Patients with neuroblastoma should have a routine clinical 123I-MIBG scintigraphy (planar and/or SPECT/CT) performed within 6 months prior to the inclusion visit or scheduled within 3 months after the inclusion visit. According to patients' condition and clinical management, part of patients with PPGL and NB will receive 68Ga-DOTATATE PET/CT, comparing with 18F-MFBG PET/CT.
  Interventions: Drug: 18F-MFBG; Drug: 68Ga-Dotatate

INTERVENTIONS:
Drug: 18F-MFBG — Patients with neuroendocrine malignancies receive 2-4 MBq/kg of 18F-MFBG intravenously followed by PET/CT after 60min of injection.
  Other Names: 18F-metafluorobenzylguanidine
Drug: 68Ga-Dotatate — Patients with malignant PPGL and NB receive intravenously 68Ga-Dotatate followed by PET/CT after 40min of injection.

SUMMARY:
The aim of this study is to evaluate the diagnostic performance and tumor burden of 18F-metafluorobenzylguanidine (18F-MFBG) positron emission tomography (PET) in patients with neuroendocrine tumors mainly in pheochromocytoma and paraganglioma (PPGL) and neuroblastoma (NB).

DETAILED DESCRIPTION:
Pheochromocytoma and paraganglioma (PPGL) and neuroblastoma (NB) highly express norepinephrine transporter (NET) which is targeted by functional analogue of norepinephrine, 131I/123I-MIBG. However, low spatial resolution of 123/131I-MIBG and inaccurate attenuation correction of single photon emission tomography (SPECT/CT) will affect the image quality of MIBG SPECT and lead to poor diagnosis of small lesions. In addition, 123I-MIBG imaging is usually performed at 24 h after injection, while 131I-MIBG is performed at 48 h or even 72 h after injection. The procedure is complicated and takes a long time, which limits clinical application. 18F-labeled MFBG is an ideal tracer to show the expression of NET. Preliminary data show that 18F-MFBG imaging is safe and has favorable biodistribution and kinetics with good targeting of lesions. Patients can undergo PET 0.5 hours after injection without special preparation. Our study will assess the safety profile, image quality and evaluate the diagnostic performance and tumor burden of 18F-MFBG on nural crest tumors including PPGL and NB. Patients with histologically confirmed or clinically suspected neural crest tumor will be prospectively recruited in this study.

ELIGIBILITY:
Inclusion Criteria:

- The subject has read, signed, and dated an informed consent form (ICF) prior to any study procedures being performed. Patients with histologically confirmed or clinically suspicious neural crest tumor.

For patients with neuroblastoma, subject should have a routine clinical 123I-MIBG scintigraphy (planar + SPECT/CT) performed within 6 months prior to the inclusion visit or scheduled within 3 months after the inclusion visit.

The subject is male or is a nonpregnant, nonlactating female who is either surgically sterile or is post-menopausal. The subject is able and willing to comply with all study procedures as described in the protocol.

Exclusion Criteria:

- Patients are potentially pregnant (serum and urinary hCG test will be performed in women where pregnancy is not excluded) or is breast-feeding.

Patients undergo surgery between the selection and inclusion visit. Patients who are pregnant, may possibly be pregnant, or wish (including their partners) to become pregnant during the study period, or are lactating. Patients who are not suitable to participate in the trial according to researchers.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The evaluation of diagnostic performance of 18F-MFBG PET in different regions in metastatic neural crest tumor. | through study completion, an average of 1 year
  Patients with histologically confirmed metastatic neural crest tumor will be prospectively recruited in this study. They will receive 18F-MFBG PETand 123I-MIBG SPECT. Rate of detected lesions (visual) in bone, lymph node and liver will be compared.

SECONDARY OUTCOMES:
Assessment of lesion targeting by 18F-MFBG as compared to 68Ga-DOTATATE | through study completion, an average of 2 years
  A lesion-by-lesion analysis will be performed to compare the number of detected lesions using 18F-MFBG and 68Ga-DOTATATE.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Li, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking union medical college hospital, Beijing, Dongcheng, China

REFERENCES:
- [Derived] Wang P, Yu S, Chen X, Zheng X, Mao J, Jing H, Zhuang H, Li F, Su X. [18F]MFBG PET/CT is an effective and preferable imaging modality for neuroblastoma in a prospective comparison with SSTR PET. Eur J Nucl Med Mol Imaging. 2026 Jan;53(2):899-909. doi: 10.1007/s00259-025-07449-y. Epub 2025 Jul 28. PMID 40717185
- [Derived] Wang P, Li T, Liu Z, Jin M, Su Y, Zhang J, Jing H, Zhuang H, Li F. [18F]MFBG PET/CT outperforming [123I]MIBG SPECT/CT in the evaluation of neuroblastoma. Eur J Nucl Med Mol Imaging. 2023 Aug;50(10):3097-3106. doi: 10.1007/s00259-023-06221-4. Epub 2023 May 9. PMID 37160439